CLINICAL TRIAL: NCT01081119
Title: Brief Voluntary Alcohol and Drug Intervention for Middle School Youth
Acronym: CHOICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AA016577 (NIH)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Alcohol Drinking; Cigarette Smoking; Marijuana Smoking
Keywords: adolescent; middle school; prevention; alcohol; cigarettes; marijuana
MeSH Terms: conditions — Alcohol Drinking; Cigarette Smoking; Marijuana Smoking; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project CHOICE (Experimental): Middle school receives Project CHOICE
  Interventions: Behavioral: Project CHOICE
- No Project CHOICE (No Intervention): Middle school does not receive Project CHOICE

INTERVENTIONS:
Behavioral: Project CHOICE — Voluntary after school program offered 1 day per week for 30 minutes
  Arms: Project CHOICE

SUMMARY:
We are currently working in 16 middle schools across Los Angeles, Santa Monica and Torrance to test out a voluntary after school program called Project CHOICE, which focuses on helping students decrease their alcohol and drug use. We are conducting surveys in all schools over three years and providing the intervention in 8 schools in the 2008-2009 school year and in the other 8 schools in the 2011-2012 school year. This is a program we have provided before in middle schools and we found that it was effective in curbing alcohol and drug use among students who voluntarily attended and among all students at the intervention school.

DETAILED DESCRIPTION:
The middle school years are peak years for initiation of alcohol and marijuana (Johnston et al., 2007). Unfortunately, most youth who engage in substance use and experience problems are unlikely to voluntarily make use of formal prevention services (D'Amico, 2005; Johnson et al., 2001; Wu et al., 2003). A small body of recent research suggests that youth may benefit from less formal programs that are brief, voluntary, and easily accessible (Brown, 2001; D'Amico et al., 2005). However, very few intervention programs of this type have been developed (Little and Harris, 2003). Thus, while this approach shows promise, the impact of intervention programs that younger teens may choose to attend has not been extensively examined. One such intervention, Project CHOICE, was developed and tested by the PI using NIAAA funding for developmental work (R21AA13284). Project CHOICE is the only voluntary intervention that has been tested for middle school youth and our small quasi-experimental study has demonstrated its efficacy in one school setting (D'Amico and Edelen, in press; D'Amico et al., 2005). The Project CHOICE intervention addresses several critical gaps in the field, including beginning to understand voluntary service utilization among this age group and assessing how this type of program may impact school-wide use of alcohol and other drugs (AOD). The main objective of the proposed 5-year longitudinal study is to build on our initial work by conducting a more rigorous test of Project CHOICE. The study will include 16 middle schools, located in the ethnically diverse Southern California cities of Los Angeles, Santa Monica, and Torrance. These schools will be randomly assigned as intervention (n= 8) or control (n = 8). We will first examine individual-level effects by testing whether Project CHOICE affects AOD-related outcomes among students who participate in the intervention. We will then examine school-level effects by testing whether AOD rates among all students in the intervention schools are affected, regardless of participation. We assume that these school-level effects will be due to changes in the school environment (e.g., Project CHOICE advertising, discussion of Project CHOICE among students, changes in social norms). In anticipation of this school-level impact, a secondary objective of this study is to gain a better understanding of who participates in Project CHOICE, as well as how these participants and changes in the school environment may influence the attitudes and behaviors of those who do not participate. This research incorporates a novel methodology for AOD involvement, as it emphasizes personal self-change efforts and natural recovery and is appealing to both using and non-using youth. The work proposed in this application represents the important next step in this line of research: to more critically evaluate Project CHOICE and its potential impact on both school-wide and individual outcomes with a larger population of youth.

ELIGIBILITY:
Inclusion Criteria: Adolescents between the ages of 11 and 15 who are currently attending one of 16 selected middle schools across Los Angeles, Torrance, and Santa Monica -

Exclusion Criteria: None

-

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6455 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Alcohol, cigarette, and marijuana use | 3 years

SECONDARY OUTCOMES:
Substance use-related cognitions | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. D'Amico, PhD, Principal Investigator — RAND
Locations (1):
- 16 middle schools in Torrance, Santa Monica, and Los Angeles, Los Angeles, California, United States